CLINICAL TRIAL: NCT02597530
Title: Effect of Different Time of Transcutaneous Electric Acupoint Stimulation(TEAS) on Acupuncture Anesthesia
Brief Title: Different Stimuli of Transcutaneous Electric Acupoint Stimulation(TEAS) on Acupuncture Anesthesia
Acronym: TEAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: wangqiang (Other)
Responsible Party: Sponsor-Investigator, wangqiang, Professor, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Xijingmazui; mazuike (Other: Xijing Hospital)
Record Dates: First submitted 2015-10-29; First posted 2015-11-05 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Acupuncture
Keywords: TEAS; anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Long-term stimulution group (Experimental): According to ancient Chinese medical books, acupoints Hegu and Zusanli are chosen and identified.Patients in Long-term stimulation group received electrical stimulation with the 'disperse-dense' waves.TEAS will be administered 30 minutes prior to anesthesia and continued until the end of the surgery with dilatational wave(2-15HZ).All patients will remove electrodes on surgery over.
  Interventions: Device: TEAS
- Short-term stimulution group (Other): According to ancient Chinese medical books, acupoints Hegu and Zusanli are chosen and identified.The patients in Short-term stimulation group received electrical stimulation with the 'disperse-dense' waves.TEAS will be administered 30 minutes prior to anesthesia and ended at time of anesthesia with dilatational wave(2-15HZ).All patients will remove electrodes on surgery over.
  Interventions: Device: TEAS
- Sham group (Placebo Comparator): Patients in sham group will be pasted electrodes 30 minutes before anesthesia but without electrical stimulation.All patients will remove electrodes on surgery over.
  Interventions: Device: TEAS

INTERVENTIONS:
Device: TEAS — According to ancient Chinese medical books, acupoints LI4,PC6 and ST36 are chosen and identified.TEAS in long-term group will be administered 30 minutes prior to anesthesia and continued until the end of the surgery. In short-term group,TEAS will be administered 30 minutes prior to anesthesia and ended at time of anesthesia.In sham group,electrodes will be pasted 30 minutes before anesthesia but without electrical stimulation.All patients will remove electrodes on surgery over.

SUMMARY:
To determine whether treating by transcutaneous electrical acupoint stimulation (TEAS) combined with general anesthetic during peri-operative could alleviate the dosage of anesthetic drugs compared with control and sham group.

DETAILED DESCRIPTION:
Acupuncture is a traditional Chinese medical technique that involves the insertion of needles at acupoints to treat diseases by Jingluo (the system of meridians, through which energy is thought to ﬂow through the body in Chinese medicine). It is usually applied to relieve pain. Several clinical trials have been conducted to evaluate the effect of electroacupuncture on the consumption of intra-operative anaesthetics and on drug-related side-effects, with promising results. Compared with acupuncture or electroacupuncture, transcutaneous electric acupoint stimulation(TEAS) is a non-invasive technique and has some advantages, including no risk of infections or needle-induced contagious disease and reduced fear of stimulation. It can potentially be applied by any anaesthetist or pre-operative personnel with minimal training.Thus, investigators conducted this controlled, prospective, double-blinded clinical trial to investigate whether treating by transcutaneous electrical acupoint stimulation combined with general anesthetic during peri-operative could alleviate the dosage of anesthetic drugs compared with control and sham group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65
2. ASA physical statusⅠorⅡ
3. Elective gynecological laparoscopic surgery under general anesthesia
4. BMI of 18 to 25
5. Duration of operation≤2 hours
6. Patient who signed the informed consent

Exclusion Criteria:

1. Pregnancy or breast-feeding women
2. Serious lung disease/Serious cardiovascular disease/Serious liver, renal abnormalities
3. Patients who have a history of gastrointestinal surgery or chronic gastrointestinal disease
4. Patient has diseases in nervous-mental system
5. Operation time more than 2 hours
6. Patients with contraindications to the use of electroacupuncture, such as skin damage or infection at the acupoints;
7. Patients with experience of transcutaneous electrical stimulation treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Consumption of remifentanil during the operation（ug/kg/min）. | intraoperative

SECONDARY OUTCOMES:
Content of endocrine hormone in the blood(angiotensin-II(ng/L),Cortisol(nmol/L),β-endorphin(ng/mL) and glucose(mmol/L)). | intraoperative
Time of extubation after operation. | intraoperative
Pain after the operation(visual analog scale (vas)). | 0 hours ,2 hours ,12 hours ,24 hours after operation
Side-effects of anesthetics(nausea,vomiting,dizziness and pruritus). | 0 hours ,2 hours ,12 hours ,24 hours after operation
Hospital stays after operation(d). | Participants will be followed for the duration of hospital stay, an expected average of 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Qiang x Qiang Wang, Study Chair — Xijing Hospital

REFERENCES:
- [Background] Wang H, Xie Y, Zhang Q, Xu N, Zhong H, Dong H, Liu L, Jiang T, Wang Q, Xiong L. Transcutaneous electric acupoint stimulation reduces intra-operative remifentanil consumption and alleviates postoperative side-effects in patients undergoing sinusotomy: a prospective, randomized, placebo-controlled trial. Br J Anaesth. 2014 Jun;112(6):1075-82. doi: 10.1093/bja/aeu001. Epub 2014 Feb 26. PMID 24576720
- [Background] Iacobone M, Citton M, Zanella S, Scarpa M, Pagura G, Tropea S, Galligioni H, Ceccherelli F, Feltracco P, Viel G, Nitti D. The effects of acupuncture after thyroid surgery: A randomized, controlled trial. Surgery. 2014 Dec;156(6):1605-12; discussion 1612-3. doi: 10.1016/j.surg.2014.08.062. Epub 2014 Nov 11. PMID 25456960
- [Background] Lee MS, Ernst E. Acupuncture for surgical conditions: an overview of systematic reviews. Int J Clin Pract. 2014 Jun;68(6):783-9. doi: 10.1111/ijcp.12372. Epub 2014 Jan 22. PMID 24447388
- [Background] Sahni N, Anand LK, Gombar K, Gombar S. Effect of intraoperative depth of anesthesia on postoperative pain and analgesic requirement: A randomized prospective observer blinded study. J Anaesthesiol Clin Pharmacol. 2011 Oct;27(4):500-5. doi: 10.4103/0970-9185.86595. PMID 22096284
- [Background] Han JS. Acupuncture analgesia: areas of consensus and controversy. Pain. 2011 Mar;152(3 Suppl):S41-S48. doi: 10.1016/j.pain.2010.10.012. No abstract available. PMID 21078546